CLINICAL TRIAL: NCT00242424
Title: Safety and Immunogenicity of Fluzone Influenza Virus Vaccine (2005-2006 Formulation) Among Healthy Children 6 to 12 Weeks of Age
Brief Title: Safety and Immunogenicity of Inactivated Influenza Virus Vaccine Among Healthy Children 6-12 Weeks of Age
Acronym: GRC28
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Janet Englund, MD, Seattle Children's Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 05065501
Record Dates: First submitted 2005-10-19; First posted 2005-10-20 (Estimated); Last update posted 2009-01-28 (Estimated); Status verified 2009-01

CONDITIONS: Inactivated Influenza Vaccine
Keywords: influenza vaccine; infants; safety; immunogenicity
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): 0.25 ml normal saline placebo given as injection to infants at 2 and 3 months of age
  Interventions: Biological: 2005-2006 trivalent inactivated influenza vaccine
- 2 (Experimental): 2005-6 Fluzone, pediatric formulation of trivalent inactivated influenza vaccine (sanofi pasteur) administered to infants at 2 and 3 months of age
  Interventions: Biological: 2005-2006 trivalent inactivated influenza vaccine

INTERVENTIONS:
Biological: 2005-2006 trivalent inactivated influenza vaccine — Children enrolled at 6-12 weeks to receive first dose, 0.25 ml of trivalent inactivated influenza vaccine, 2005-6 pediatric Fluzone formulation (sanofi pastuer), with concomitant routine pediatric vaccines. Second dose administered 4 weeks later.

SUMMARY:
Study of the safety and immunogenicity (antibody producing capability) comparing inactivated influenza vaccine to placebo given to infants at 2 and 3 months of age. Infants will receive inactivated influenza vaccine at the same time as other vaccines on the routine immunization schedule. Infants will be randomized at enrollment to receive inactivated influenza vaccine or placebo at a 2:1 ratio. This study is double-blind, randomized, and placebo-controlled.

DETAILED DESCRIPTION:
Methods: A double-blind, randomized, placebo-controlled trial was conducted in 1375 healthy US infants 6-12 weeks of age. Subjects received either 2 doses of trivalent inactivated influenza vaccine (TIV, Fluzone®, sanofi pasteur 2005-6 pediatric formulation) (N=915) or placebo (N=460) 1 month apart, along with indicated concomitant vaccines. Solicited adverse events were collected for 7 days following each vaccination, unsolicited adverse events for 28 days, and serious adverse events for 6 months. Hemagglutination inhibition antibodies to all 3 vaccine strains were measured following the second TIV/placebo dose.

Results: No significant differences were seen between TIV and placebo groups for any safety outcomes. Fever ≥38oC rectal within 3 days of vaccination was seen in 11.2% vs 11.7% of TIV vs placebo recipients. Serious adverse events within 28 days of vaccine/placebo were reported in 1.9% of TIV and 1.5% of placebo recipients; only one (hypersensitivity reaction in a TIV recipient) was considered vaccine-related. Significantly increased antibody responses (p<0.001) were seen against all 3 strains in TIV recipients by titer ≥ 1:40 or geometric mean titer (GMT) (p<0.001). Altogether, 50% of infants had antibody titers ≥ 1:40 for H1N1, 86% for H3N2, and 11% for B compared with 7%, 10%, and 0.3% in the placebo group. The reciprocal GMT for influenza recipients was 33, 95, and 11 for H1N1, H3N2, and B vs. 7, 9, and 5 for placebo recipients. Over 90% of infants who received TIV had antibody ≥ 1:40 for at least one vaccine strain and 49.6% for 2 strains, vs. 16.4% and 0.9% in the placebo group.

Conclusions: TIV administered to young infants beginning at 6-12 weeks of age is safe and immunogenic.

ELIGIBILITY:
Inclusion Criteria:

* Age 42 to 84 days on the day of inclusion
* Full term (born at >=36 weeks with birth weight >=2.5 kg
* Considered to be in good health
* Parental consent obtained and available
* Available for the study duration (6 months)

Exclusion Criteria:

* Reported allergy to egg proteins, chicken proteins
* Previous history of influenza vaccination or disease
* Receipt of any vaccine other than Hepatitis B prior to enrollment
* Acute illness with rectal temperature >= 38.0 (defer enrollment)
* Known bleeding disorder
* Participation in other interventional clinical trial within 30 days prior to enrollment

Ages: 42 Days to 84 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1375 (Actual)
Dates: Start 2005-09; Primary Completion 2006-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
To demonstrate the safety of Fluzone vaccine administered to 2-month old children | within 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Janet A Englund, MD, Study Chair — Seattle Children's Hospital
Locations (1):
- Seattle Children's Hospital and Regional Medical Center, Seattle, Washington, United States

REFERENCES:
- [Result] Englund JA, Walter EB, Black S, et al. Safety and Immunogenicity of Fluzone Trivalent Inactivated Influenza Vaccine (TIV) in Infants 6-12 Weeks of Age. Presented at Infectious Disease Society of America (IDSA), Toronto, Oct. 14, 2006